CLINICAL TRIAL: NCT05865197
Title: Feasibility of Home-based, Ambient Passive Sensor Technology to Provide Early Warning of Health Decompensation by Detecting Deviations in Activities of Daily Living (ADLs) of Elderly Subjects With Diagnosed Chronic Heart Failure
Brief Title: Evaluation of Home-based Sensor System to Detect Health Decompensation in Elderly Patients With History of CHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sensorum Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Sensorum P-002
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: CHF; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Passive monitoring: No intervention
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection of clinically relevant signals using home-based sensor system

SUMMARY:
Sensorum Health (Sensorum) is conducting a pilot study to determine if Sensorum's proprietary passive sensor network can be used to identify signals of early health decompensation in subjects prior to a hospitalization for chronic disease exacerbation or other ambulatory care sensitive conditions. Successful early detection would provide a window of opportunity to intervene outside of the acute setting in future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Current Patient at Weill Cornell Medicine
* Aged 55 years or older
* Able to consent
* Documented diagnosis of congestive heart failure (CHF)
* At least 1 of the following prior hospital utilization events in the past 12 months
* Inpatient admission for any reason
* Facility observation stay for any reason
* Emergency Department visit for any reason

Exclusion Criteria:

* Significant cardiac valvular disease
* End-Stage Renal Disease (ESRD)
* End-Stage CHF
* End-Stage COPD

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current Patient of PI's clinic at Weill Cornell Medicine
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Recall of AI in passive sensor system | 6 months
  Evaluation of AI ability to prospectively detect hospital utilization event
Precision of AI in passive sensor system | 6 months
  Evaluation of AI ability to precisely predict hospital utilization event

SECONDARY OUTCOMES:
Recall of sensor data review by trained nurses | 6 months
  Evaluation of nurse ability to prospectively detect hospital utilization event
Precision of sensor data review by trained nurses | 6 months
  Evaluation of nurse ability to precisely predict hospital utilization event

CONTACTS AND LOCATIONS:
Overall Officials: Parag Goyal, M.D., MSc, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No